CLINICAL TRIAL: NCT07018206
Title: Impact Of Upadacitinib On The Frequency Of Acute Recurrent Anterior Uveitis In Patients With Axial Spondyloarthritis (UP-FOR-U)
Brief Title: Impact Of Upadacitinib On The Frequency Of Acute Recurrent Anterior Uveitis In Patients With Axial Spondyloarthritis
Acronym: UP-FOR-U
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CARE ARTHRITIS LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B25-723
Record Dates: First submitted 2025-05-27; First posted 2025-06-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Axial Spondylarthritis (axSpA)
Keywords: Axial Spondyloarthritis; Acute Anterior Uveitis
MeSH Terms: conditions — Axial Spondyloarthritis; Uveitis, Anterior | interventions — upadacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Upadacitinib (Experimental): All participants enrolled in the study will receive 15 mg of Upadacitinib per day for 52 weeks.
  Interventions: Drug: Upadacitinib 15 MG [Rinvoq]

INTERVENTIONS:
Drug: Upadacitinib 15 MG [Rinvoq] — 15mg tablet once per day

SUMMARY:
This is a Phase IV, open-label, multicenter study evaluating the impact of upadacitinib on the frequency of acute anterior uveitis (AAU) in adults with axial spondyloarthritis (axSpA) and a documented history of AAU in the prior 52 weeks. Approximately 200 participants will be enrolled across North America and Europe, including both biologic DMARD-inadequate responders (bDMARD-IR) and bDMARD-naïve patients. The primary objective is to assess the change in exposure-adjusted AAU event rate during 52 weeks of treatment with upadacitinib 15 mg once daily. Secondary objectives include evaluating the effect of upadacitinib on disease activity, pain, physical function, quality of life, and sleep. Safety and tolerability will also be assessed throughout the study.

DETAILED DESCRIPTION:
The UP-FOR-U study is a Phase IV, open-label, interventional study designed to assess the effect of upadacitinib 15 mg once daily on the frequency of acute anterior uveitis (AAU) in adult patients with axial spondyloarthritis (axSpA) and a history of ophthalmologist-confirmed AAU in the 52 weeks prior to baseline. The study will enroll approximately 200 participants across 20 sites in Canada, the United States, and the European Union, comprising both biologic DMARD-inadequate responders (bDMARD-IR) and bDMARD-naïve patients. All participants will receive open-label treatment with upadacitinib for 52 weeks, with monthly remote visits and quarterly in-person visits.

The primary objective is to evaluate the change in the exposure-adjusted incidence rate of ophthalmologist-confirmed AAU events per 100 patient-years during treatment, compared to the 52-week pre-study period. Secondary outcomes include measures of disease activity (e.g., ASDAS), physical function (e.g., BASFI), quality of life (e.g., ASAS-HI, SF-12), pain, sleep (e.g., PSQI), and safety (including adverse events, adverse events of special interest, and serious adverse events).

This study reflects real-world clinical practice and incorporates remote data collection and patient-reported outcomes to improve feasibility and patient engagement. It is designed in accordance with ICH-GCP, FDA, Health Canada, and EMA regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Subject ≥18 of age at the screening visit.
2. Subject must be able to understand and willing to adhere to all protocol requirements and voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.
3. Diagnosis of axSpA by their treating rheumatologist.
4. Classification of axSpA according to ASAS Classification Criteria
5. History of at least one acute anterior uveitis event in the 52 week period prior to baseline, diagnosed by an ophthalmologist.
6. Active disease as defined by a BASDAI value of ≥4 and TBP score of ≥4 (on a 0-10 NRS scale) at screening and baseline.
7. History of an inadequate response to at least two different NSAIDs over a period of 4 weeks in total at the maximum recommended or tolerated doses, or intolerance/contraindication (e.g., allergic reaction, gastrointestinal symptoms or signs, severe arterial hypertension, etc.) for NSAIDs.
8. Subjects must have been treated for ≥3 consecutive months prior to the study entry with bDMARD therapy and/or for ≥4 weeks of NSAID therapy, in accordance with local product label for AS or nr-axSpA, but continue to exhibit active SpA, or had to discontinue previous bDMARD and/or NSAID treatment due to intolerability or toxicity, irrespective of treatment duration. A total of 50 subjects who are bDMARD-naïve and 150 subjects who are b-DMARD-IR will be included in the study.
9. For all females of child-bearing potential: must not have a positive serum pregnancy test at the Screening Visit and must have a negative urine pregnancy test at Baseline prior to the first dose of study drug (local practices may require serum pregnancy testing at Baseline). Subjects with a borderline serum pregnancy test at Screening must have absence of clinical suspicion of pregnancy or other pathological causes of borderline results and a serum pregnancy test ≥3 days later to document continued lack of a positive result (unless prohibited by local requirements).
10. Subjects who are regularly taking NSAIDs or analgesics (including low potency opioids) as part of their axSpA therapy are required to be on a stable dose/dose regimen for at least 7 days prior to the baseline visit. If entering the study on concomitant tramadol, combination of acetaminophen/paracetamol and codeine or combination of acetaminophen/paracetamol and hydrocodone, and/or non-opioid analgesics, subject must be on stable dose(s) for at least 7 days prior to the baseline Visit. However, subject must not have used opioid analgesics (except for combination of acetaminophen/paracetamol and codeine or combination of acetaminophen/paracetamol and hydrocodone which are allowed) within 7 days prior to the BL Visit.
11. Subjects taking oral corticosteroids must be on an average daily and stable dose of ≤10mg/day prednisone or equivalent for at least 14 days prior to the baseline visit.
12. Subjects entering the study on the following concomitant csDMARDs must be on a stable dose as indicated below for at least 28 days prior to the baseline Visit (in case of Leflunomide washout must be either 11 days with colestyramine or 30 days with activated charcoal or as per local label). A combination of up to 2 background csDMARDs is allowed EXCEPT the combination of methotrexate (MTX) and leflunomide. • MTX (≤ 25 mg/week); or • Sulfasalazine (SSZ) (≤ 3 g/day); or • Hydroxychloroquine (≤ 400 mg/day); or • Chloroquine (≤ 250 mg/day); or • Leflunomide (≤ 20 mg/day)
13. If subjects are currently taking bDMARD therapy, they may be recruited after an appropriate wash-out period of bDMARD prior to the Baseline Visit. Washout periods are as follows: 4 weeks for Etanercept, 8 weeks for Infliximab, Golimumab, and Certolizumab, 10 weeks for Adalimumab, and Ixekizumab, 12 weeks for Secukinumab. However, subjects should not stop their previous successful biological therapy only to be included in this study. For subjects intolerant to bDMARD and not on such treatment a washout period may not be necessary.

Exclusion Criteria:

1. Active infection(s) requiring treatment with parenteral anti-infectives within 30 days, or oral antiinfectives within 14 days prior to the baseline Visit; Chronic recurring infection and/or active viral infection that based on the investigator's clinical assessment makes the subject an unsuitable candidate for the study.
2. COVID-19: In subjects who tested positive for COVID-19, at least 5 days must have passed between a COVID-19 positive test result and the Baseline visit of asymptomatic subjects. Subjects with mild/moderate COVID-19 infection can be enrolled if fever is resolved without use of antipyretics for 24 hours and other symptoms improved, or if 5 days have passed since the COVID-19 positive test result (whichever comes last). Subjects may be rescreened if deemed appropriate by the investigator based upon the subject's health status
3. Suspected COVID-19: subjects with signs/symptoms suggestive of COVID-19, known exposure, or high-risk behavior should undergo molecular (e.g., PCR) testing to rule out SARS-CoV-2 infection or must be asymptomatic for 5 days from a potential exposure;
4. History of recurrent (more than one episode) herpes zoster or disseminated/multi-dermatomal (a single episode) herpes zoster or disseminated (a single episode) herpes simplex.
5. Primary or secondary immunodeficiency.
6. Subjects with active TB or who meet TB exclusionary parameters (specific requirements for TB testing are provided in Section 7.0: TB Testing/TB Prophylaxis)
7. Chronic infection with hepatitis B virus. At screening HBsAg and anti-HBc will be tested. Subjects who are HBsAg positive will be excluded. In case of HBsAg negativity, but anti-HBc positivity, participation in the study is possible if HBV-DNA testing is negative and no exclusionary liver function tests.
8. Chronic infection with hepatitis C (HCV) (HCV ribonucleic acid (RNA) detectable in any subject with anti-HCV antibody (HCV Ab), or Human Immunodeficiency Virus (HIV) infection confirmed by positive HIV-antibody and antigen test.
9. Female subjects who are breastfeeding, pregnant, or plan to become pregnant during the study or within 4 weeks following the last dose of study drug.
10. Subjects with chronic inflammatory articular disease (other than axSpA or systemic autoimmune diseases, e.g., systemic lupus erythematosus, Sjögren´s syndrome, RA, unequivocal chronic fatigue syndrome, or unequivocal fibromyalgia. Subjects with a diagnosis of Crohn's disease or ulcerative colitis are allowed as long as they have no active symptomatic disease within 4 weeks prior to BL.
11. Concomitant treatment with strong inductors or inhibitors of cytochrome P450 3A (e.g., Ketoconazole, Fluconazole, Rifampicin, Clarithromycin, St-John´s-wort).
12. Prior treatment with upadacitinib or another JAK-inhibitor or TYK2-inhibitor for axSpA.
13. History of hypersensitivity to any component of upadacitinib tablets.
14. Treatment with intravenous, intramuscular or intraarticular/periarticular, or intrarectal steroids within 4 weeks prior to baseline Visit; treatment with oral steroids in a dose of >10 mg prednisolone equivalent per day within 4 weeks prior to baseline visit.
15. Subject must not have been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or five half-lives (whichever is longer) prior to the first dose of study drug or is currently enrolled in another interventional clinical study.
16. History of an infected joint prosthesis at any time, with the prosthesis still in situ.
17. Actual malignancies or history of malignancies with curative treatment within 5 years prior to screening, except successfully treated non-metastatic squamous cell or basal cell carcinoma of the cutis or carcinoma in situ of the cervix.
18. A subject with any condition possibly affecting oral drug absorption, e.g., gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery such as gastric bypass. Procedures such as gastric banding, that simply divides the stomach into separate chambers, are NOT exclusionary.
19. Significant trauma or surgery procedure within 4 weeks prior to baseline.
20. Evidence of other severe uncontrolled gastrointestinal, hepatic (serum albumin <25 mg/l or ChildPugh-Score >10), renal, pulmonary, cardiovascular, nervous or endocrine disorders.
21. Any history of prior cardiovascular event, including but not limited to cerebrovascular accident, myocardial infarction, coronary stenting, and aorto-coronary bypass surgery.
22. History of thrombosis and/or hematological disorder increasing the propensity to thrombosis.
23. Any subject who has been vaccinated with live or attenuated vaccines within the 4 weeks prior to the first dose of study medication or is to be vaccinated with these vaccines at any time during treatment or within 4 weeks after the last dose of study drug.
24. Any of the following lab abnormalities detected at screening: a) Hemoglobin <9 g/dl; b) Absolute neutrophil count (ANC) <1.2 x 109/L (<1020/mm3) c) Absolute lymphocyte count (ALC) <0.750 x 109/L (<750/mm3) d) Platelet count <9 g/dL e) Liver function tests (LFT) >2 x ULN f) Serum apartate transaminase (AST) >2 x ULN g) Serum alanine transaminase (ALT) >2 x ULN; h) Estimated glomerular filtration rate (GFR) by simplified 4-variable MDRD formula < 30 mL/min/1.73 m2; i) Total white blood cell (WBC) count < 2,500/μL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of recurrent acute anterior uveitis (AAU) | 52 Weeks
  To evaluate the impact of upadacitinib on the frequency of recurrent acute anterior uveitis (AAU) over 52 weeks in subjects with active axSpA and a prior AAU event in the 52 weeks prior to baseline, who are switching from bDMARD (North America and Europe), or who are NSAID-IR and bDMARD naïve (Europe), in real world practice.

SECONDARY OUTCOMES:
Proportion of participants achieving low disease activity (ASDAS LDA) at Week 24 | Week 24
  The percentage of participants achieving a score of less than 2.1 on the Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 24. ASDAS is a validated composite index that incorporates patient-reported outcomes and objective measures of inflammation to assess disease activity in axial spondyloarthritis.
Proportion of participants achieving ASAS Health Index (ASAS-HI) ≤5 at Week 52 | Week 52
  The percentage of participants who achieve a score of 5 or less on the ASAS Health Index (ASAS-HI) at Week 52. The ASAS-HI is a validated patient-reported outcome measure that evaluates the impact of axial spondyloarthritis on physical function, pain, emotional well-being, and social participation. A score ≤5 indicates better health status and is considered a meaningful clinical threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Maksymowych, Dr., Principal Investigator — CARE ARTHRITIS LTD.
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided